CLINICAL TRIAL: NCT04925895
Title: Dynamic Soft Tissue Mobilization vs Proprioceptive Neuromuscular Facilitation in Reducing Hamstring Muscle Tightness in Patients With Knee Osteoarthritis: a Randomized Control Trial
Brief Title: Effects of Dynamic Soft Tissue Mobilization in Reducing Hamstring Tightness in Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Syed Shahzad Ali, Principal Investigator, Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00003
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Knee Osteoarthritis; Muscle Tightness; Range of Motion; Dynamic Stretching
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Muscle Stretching Exercises; Cryotherapy; Exercise

STUDY DESIGN:
Intervention Model Description: A single blinded randomized control trial in which total 48 patients will be enrolled and randomly allocated into 2 interventional groups equally. The randomization will be carried out through an open source software "research randomizer" by statistician.
Who Masked: Outcomes Assessor
Masking Description: Other than the principal investigator, another physiotherapist will work as outcomes assessor who will blind to the intervention type given to the patient who will be assessed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dynamic soft tissue mobilization (Experimental): Dynamic soft tissue mobilization (DSTM) is a soft tissue mobilization technique use to treat tight spasm using progressive muscle activation.
  Interventions: Other: Dynamic soft tissue mobilization; Other: Cryotherapy; Other: Isometric knee strengthening excercises
- Proprioceptive neuromuscular facilitation stretching (Active Comparator): PNF stretching technique, a type of flexibility training that is effective in improving muscle flexibility and restore functional ranges using a wide array of techniques.
  Interventions: Other: Proprioceptive neuromuscular facilitation stretching; Other: Cryotherapy; Other: Isometric knee strengthening excercises

INTERVENTIONS:
Other: Dynamic soft tissue mobilization — Dynamic soft tissue mobilization will be given in the following sequence, In supine position with 90˚ flexion of knee and hip joint deep longitudinal strokes will be applied from distal to proximal direction along with the tightened area of hamstring while passively stretching the hamstring. Total 5 longitudinal strokes will be applied followed by shaking for 20 seconds. Then progressed to the next dynamic technique in the above-mentioned sequence but the patient will be asked to do leg extension actively to achieve reciprocal inhibition of the hamstring muscle. In The next step, the subject will apply a force to the therapist's hand to engage the hamstring eccentrically as the muscle will be lengthened to its end range. In that position, the therapist will apply 5 deep longitudinal strokes from the distal towards the proximal direction on tight hamstring muscles.
  Other Names: DSTM; dynamic soft tissue technique; soft tissue mobilization
  Arms: Dynamic soft tissue mobilization
Other: Proprioceptive neuromuscular facilitation stretching — The position of the patient will be supine lying with 90⁰ flexion of hip. Therapist will passively extend the knee joint where patient will feel a mild stretch. Then therapist will ask the patient to do knee flexion in counter resistance applied by the therapist by using about 50% of his maximum strength and isometric contraction of hamstring muscles will be achieved. Patient will maintain that isometric contraction for 8 seconds then relax on therapist command. Just after relaxation therapist will further stretch the hamstring muscle to the point of mild to moderate painless stretch and patient will hold it for 30 seconds. Three repetitions will be applied in each session.
  Other Names: PNF stretchings; PNF exercises; PNF stretching exercise
  Arms: Proprioceptive neuromuscular facilitation stretching
Other: Cryotherapy — application of cold pack on knee joint for 10 minutes
  Other Names: Cold pack; Icing
Other: Isometric knee strengthening excercises — i. Isometric hip adductors exercises in crook lying: Two sets of 10 repetitions with a 10-seconds hold will be carried out.
  ii. Isometric quadriceps strengthening exercises in supine lying: A towel roll underneath the knee joint will be used to perform this exercise. Two sets of 10 repetitions with a 10-seconds hold will be performed.
  Other Names: Isometrics; knee strengthening exercises; Isometric quads

SUMMARY:
The objective of this randomized control trial is to evaluate the effectiveness of dynamic soft tissue mobilization in comparison with the proprioceptive neuromuscular facilitation (hold-relax) technique in reducing hamstring muscle tightness, pain and improving physical functions in patients with knee osteoarthritis by using Visual Analog Scale-10 cm, Active Knee Extension Angle Test in degree and Knee Injury and Osteoarthritis Outcome Score. This study will be carried out at Sindh Institute of Physical Medicine and Rehabilitation and Dow Institute of Physical Medicine and Rehabilitation, Dow University of Health Sciences, Karachi on the basis of non-probability purposive sample technique with screening for study criteria through a consultant physician (blinded) . After taking informed consent all participants will be randomly allocated into 2 groups i.e. 24 in interventional group 'A' and 24 in interventional group 'B' through second researcher who is not involved in screening, baseline assessment and providing intervention.The interventional group 'A' will received dynamic soft tissue mobilization on hamstring muscle along with cryotherapy on knee joint and isometric strengthening exercises for knee osteoarthritis while the interventional group 'B' will received proprioceptive neuromuscular facilitation (hold relax) technique on hamstring muscle along with cryotherapy on knee joint and isometric strengthening exercises for knee osteoarthritis. Twelve sessions will be given each of 30 minutes.Outcomes will be assessed at baseline and at last session.

DETAILED DESCRIPTION:
All the participants will referred by the physiatrist as diagnosed with knee osteoarthritis. All the data will be collected within ethical constraints. Only principal investigator will access to the data as it will be in her custody. Patient recruitment, data collection, data management, data analysis, reporting for adverse events, and change management will be strictly performed within codes of ethics.

The sample size of 48 patients (24 in one group) is calculated by using open epi software version 3, Paired Means Power Analysis with 99% Confidence Interval and 95% power of test, mean ± S.D of VAS 5.27 ± 0.8 in group A and 3.81±1.4 in group B on the basis of previous findings. The missing data will be considered during analysis and results interpretation for any inconsistency in results.Data were stored and analyzed using IBM-SPSS version 23.0, Mean with standard deviation will be calculated for all quantitative variables. Counts with percentages will be presented for quantitative variables. parametric or non parametric tests will be used to compare outcome variables within and between groups after sessions completion. P-values less than 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Both genders
* Subjects with 40 years of age and above
* Patients with hamstring tightness
* ACR clinical + radiological classification criteria for knee osteoarthritis

Exclusion Criteria:

* Patients with positive sciatic nerve test (SLR)
* Patients with neurological disorder impacting on lower extremity
* Musculoskeletal knee deformity e.g. varus
* Patients with lower limb internal fixation
* History of previous lower limb arthroplasty or another knee surgery
* Patients with history of infectious disease or malignancy effecting the lower extremity .
* Using assistive device(stick/cane)
* History of spinal surgery
* Patient having low backache or sciatica

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-04-22 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-10 (Actual)

PRIMARY OUTCOMES:
Visual analogue scale in centimetre | upto 4 weeks
  A bidirectional scale for subjective measurement for pain comprises of a 10 cm line labeling parallel on both sides, starts with least "no pain" (0 cm) and end on most "worst pain" (10 cm).
Active Knee Extension Angle Test in degree | upto 4 weeks
  It will used to assessing the hamstring muscle length by using goniometry with 90° of hip flexion. higher the degree higher will be the knee extension.

SECONDARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score | upto 4 weeks
  It is a patient related outcome measure, having 5 sub-scales, designed to check disease development and outcomes followed by surgical, pharmaceutical, physical therapy or other interventions.100 indicates no problem and 0 indicates extreme problem.

CONTACTS AND LOCATIONS:
Overall Officials: Khadija Nafees, MSAPT, Principal Investigator — Dow University of Health Sciences; Shahzad Ali Syed, MSPT, Study Chair — Dow University of Health Sciences; Aftab Ahmed Mirza Baig, MSAPT, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Nafees K, Baig AAM, Ali SS, Ishaque F. Dynamic soft tissue mobilization versus proprioceptive neuromuscular facilitation in reducing hamstring muscle tightness in patients with knee osteoarthritis: a randomized control trial. BMC Musculoskelet Disord. 2023 Jun 2;24(1):447. doi: 10.1186/s12891-023-06571-y. PMID 37268961